CLINICAL TRIAL: NCT05472623
Title: Phase 2 Trial of Neoadjuvant KRAS G12C Directed Therapy With Adagrasib (MRTX849) With or Without Nivolumab in Resectable Non-Small Cell Lung Cancer (Neo-KAN)
Brief Title: Neoadjuvant KRAS G12C Directed Therapy With Adagrasib (MRTX849) With or Without Nivolumab
Acronym: Neo-Kan
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no participants enrolled across sites
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Mirati Therapeutics Inc. (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB00306149
Record Dates: First submitted 2022-07-21; First posted 2022-07-25 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Resectable Non-Small Cell Lung Cancer
Keywords: Adagrasib; Nivolumab; Neoadjuvant; Resectable; NSCLC
MeSH Terms: interventions — adagrasib; Nivolumab

STUDY DESIGN:
Intervention Model Description: The study will enroll patients with newly diagnosed, biopsy-proven stage IB-IIIA NSCLC deemed surgically resectable and fit for surgery by a multidisciplinary thoracic oncology team. The study will accrue 42 patients to the following two arms sequentially:
  * Arm A: oral Adagrasib 600 mg twice daily for 6 weeks prior to surgery (21 patients)
  * Arm B: oral Adagrasib 400 mg twice daily for 6 weeks and IV nivolumab 240 mg every 2 weeks for 3 doses prior to surgery (21 patients)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Active Comparator): Arm A treatment: Oral Adagrasib 600 mg twice daily for 6 weeks prior to surgery. Surgical Resection, then standard postoperative therapy(chemo +/- RT).
  Interventions: Drug: Adagrasib
- Arm B (Active Comparator): Arm B treatment: Oral Adagrasib 400 mg twice daily for 6 weeks and IV Nivolumab 240mg every 2 weeks for 3 doses prior to surgery. Surgical Resection, then standard postoperative therapy(chemo +/- RT).
  Interventions: Combination Product: Adagrasib/Nivolumab

INTERVENTIONS:
Drug: Adagrasib — Oral Adagrasib 600 mg twice daily for 6 weeks prior to surgery.
  Arms: Arm A
Combination Product: Adagrasib/Nivolumab — Oral Adagrasib 400 mg twice daily for 6 weeks and IV nivolumab 240mg every 2 weeks for 3 doses prior to surgery.
  Arms: Arm B

SUMMARY:
This is an open label phase 2 clinical trial evaluating the clinical safety, feasibility and efficacy of neoadjuvant Adagrasib alone or in combination with nivolumab in patients with NSCLC with KRAS G12C mutation.

DETAILED DESCRIPTION:
Approximately 30% of patients with non-small cell lung cancer (NSCLC) present with resectable disease, but following surgery, the majority will experience relapse and death from the cancer. Despite significant advances in therapy for advanced NSCLC, no new systemic neoadjuvant therapies have been approved for resectable NSCLC without an EGFR driver mutation in over 15 years, and these patients are in critical need of new treatments to improve rates of cure. Currently, the standard approach for resectable stage II and III disease is 3-4 cycles of pre- or postoperative chemotherapy, which provides an absolute 5-year survival benefit of only 5% over surgery alone.

Neoadjuvant systemic therapy provides an opportunity to improve outcomes with surgery at a similar rate to adjuvant therapy, and is a more useful platform for advancing the development of new targeted and combination therapies. Pathologic complete response (pCR) and major pathologic response (MPR, ≤10% residual viable tumor) in the resected specimen serve as surrogate endpoints for event-free and overall survival, and are useful early efficacy endpoints to accelerate drug development. In resectable NSCLC, the rates of pCR and MPR with neoadjuvant immunotherapy alone are about 10% and 45% as compared to 4% and 20% with current standard of care chemotherapy. The recent approval of osimertinib in resected EGFR-mutated NSCLC has demonstrated the efficacy of targeted therapy in resectable disease, but is only available to a small minority of NSCLC patients.

KRAS is the most commonly mutated oncogene in cancer representing a vast unmet clinical need, particularly in NSCLC where it is associated with smoking history and mutated in 30% of lung adenocarcinomas. Activating KRAS mutations promote signaling pathways for growth, survival and differentiation. The most common mutant allele is KRAS G12C, present in 1 in 8 patients with NSCLC (12.5%), and represents an aggressive NSCLC phenotype with significantly higher risk of recurrence following resection in stage I-III disease.

Adagrasib is a novel small molecule inhibitor of KRAS G12C producing potent inhibition of KRAS-dependent signal transduction with high selectivity. Adagrasib has shown promise in advanced NSCLC, with 45% confirmed objective response rate and 96% disease control rate in the phase 1/2 KRYSTAL study.

Finally, the investigators anticipate enhanced efficacy of Adagrasib in combination with immune checkpoint blockade. Emerging clinical data suggests that Adagrasib reconditions the tumor immune microenvironment to become more immune-sensitive (e.g. in immune "cold" STK11 co-mutated tumors), and combination treatment with anti-PD-1 therapy resulted in increased durable responses compared to either agent alone in a murine model. Adagrasib is well-tolerated and has been safely combined with anti-PD1 therapy in a phase I trial. This will be the first study to bring this combination forward in resectable lung cancer.

This phase 2 clinical trial investigates the role of targeted KRAS G12C inhibition with and without the anti-PD-1 agent nivolumab in resectable NSCLC

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histologically confirmed diagnosis of NSCLC (squamous or nonsquamous) with KRAS G12C mutation.

  * Diagnostic core biopsy specimens must be reviewed by a faculty pathologist at the enrolling/treating institution, and biopsy tissue must be available for further biomarker evaluation. If no archived tissue is available, patients will require a repeat biopsy prior to initiation of study treatment. See section 6.5.1 and lab manual for details of pretreatment biopsy tissue required.
  * KRAS G12C mutation determined by any CLIA-certified testing platform on patient tumor tissue or plasma sample.
* Stage IB-IIIA NSCLC

  * T2aN0, T3N0, T1-2N1, T3-4N1, T1-2N2. This includes T2aN0 tumors ≥3 cm. Subjects with N3 nodal involvement are not included.
* Primary resection option for potential cure as assessed by a faculty surgeon at treating institution.
* ECOG performance status 0-1 (See Appendix B)
* Adequate organ function within the screening period as follows:

  * Leukocytes ≥ 2,000/mm3
  * Absolute neutrophil count (ANC) ≥ 1000/mm3
  * Platelet count ≥ 100,000/mm3
  * Hemoglobin ≥ 9 g/dL
  * Creatinine ≤ 1.5 x institutional upper limit of normal (ULN) or creatinine clearance (CrCl) ≥60 mL/min
  * Total Bilirubin ≤ 1.5 x institutional ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
  * AST(SGOT), ALT(SGPT), and alkaline phosphatase ≤ 3 x institutional ULN
* Pulmonary Function Testing to include DLCO must be performed to determine feasibility of surgical resection.
* Women of child-bearing potential (WOCBP):

  * Agree to use contraception while participating in this study, and for a period of 6 months following last dose of Adagrasib or nivolumab, as effects of these agents on the developing human fetus are unknown. Men whose partner is a WOCBP must also agree to use contraception during this period.
  * Negative pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within two weeks of registration.
  * Women must not be breastfeeding or plan to breastfeed for the duration of therapy or 6 months after.
* Completed informed consent process, including signing IRB/EC-approved informed consent form.
* Willing and able to comply with clinical trial instructions and requirements. Subjects must be competent to report AEs, understand the drug dosing schedule, and use of medications to control AEs.

Exclusion Criteria:

* Patients presenting with any of the following will not be included in the study:

  * NSCLC not amenable to curative intent resection based on evaluation by faculty surgeon at treating institution.

    * This includes any patient with pathologically confirmed N3 disease.
  * Prior systemic treatment for lung cancer including chemotherapy, immune checkpoint inhibitor therapy, or a therapy targeting KRAS G12C mutation.
  * Prior thoracic radiation.
  * Any concurrent malignancies for which active therapy is being received.

    * Exceptions: non-melanoma skin cancers; in situ dysplasia of the bladder, gastric, breast, colon, or cervix
  * Brain metastases at time of screening.

    * All patients must have brain imaging prior to enrollment (MRI brain or CT brain with contrast preferred).
  * Active or prior documented autoimmune or inflammatory disease as follows (Arm B only):

    * Medically relevant autoimmune disease requiring systemic treatment within 2 years prior to the first dose of study treatment.
  * Systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration (Arm B only). Inhaled or topical steroids are permitted.

    * Adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
  * Major surgery within 4 weeks prior to first dose of study treatment.
  * History of allogeneic transplant or primary immunodeficiency.
  * Uncontrolled human immunodeficiency virus (HIV) infection or acute or chronic hepatitis B or C infection.

    * Patients treated for hepatitis C with no detectable viral load and patients treated for HIV with no detectable viral load for at least 1 month while on a stable regimen of agents that are not strong inhibitors of CYP3A4 are permitted.
    * HIV testing is not required in absence of clinical suspicion of HIV.
  * Any of the following cardiac abnormalities:

    * Unstable angina pectoris or myocardial infarction within the past 6 months.
    * Symptomatic or uncontrolled atrial fibrillation within the past 6 months.
    * Congestive heart failure ≥NYHA Class 3 within the past 6 months.
    * QTc ≥ 480 msec in screening ECG measured using standard institutional method or history of familial long QT syndrome.
  * Ongoing need for a medication with any of the following characteristics that cannot be switched to alternative treatment prior to study entry (see Appendix D): known risk of Torsades de Pointes; substrate of CYP3A with narrow therapeutic index; strong inducer or inhibitor of CYP3A and/or P-gp; strong inhibitor of BCRP; and proton pump inhibitors.
  * History of stroke or transient ischemic attack within 6 months prior to first dose of study treatment.
  * History of intestinal disease or major gastric surgery likely to alter absorption of study treatment or inability to swallow oral medications.
  * Underlying medical conditions that, in the Investigator's opinion, will make the administration of study drug hazardous or obscure the interpretation of toxicity or adverse events.
  * Women who are pregnant or nursing.
  * Prisoners or subjects who are involuntarily incarcerated or compulsorily detained for treatment of either a psychiatric or physical (e.g. infectious disease) illness.
  * Receipt of a live vaccine within 30 days prior to first dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Pathologic complete response (pCR) rate | Within 90 days of surgery
  Number of patients with absence of any residual viable tumor (0%) as determined by pathologic review of surgical resection specimens divided by total number of patients in each arm started on investigational therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Marrone, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No